CLINICAL TRIAL: NCT00276705
Title: Hepatocellular Carcinoma Family of Tumours In Children / Adolescents and Young Adults
Brief Title: Combination Chemotherapy and Thalidomide in Treating Younger Patients Undergoing Surgery For Newly Diagnosed Liver Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Children's Cancer and Leukaemia Group (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000454579; CCLG-LT-2005-05; CCLG-SIOPEL-HCC; CCLG-SIOPEL-5; EU-20590; EUDRACT-2005-000427-42
Record Dates: First submitted 2006-01-12; First posted 2006-01-13 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2009-06

CONDITIONS: Liver Cancer
Keywords: adult primary hepatocellular carcinoma; childhood hepatocellular carcinoma; advanced adult primary liver cancer; localized resectable adult primary liver cancer; localized unresectable adult primary liver cancer; stage I childhood liver cancer; stage II childhood liver cancer; stage III childhood liver cancer; stage IV childhood liver cancer
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular | interventions — Cisplatin; Cyclophosphamide; Doxorubicin; Thalidomide; Chemotherapy, Adjuvant; Neoadjuvant Therapy

INTERVENTIONS:
Drug: cisplatin
Drug: cyclophosphamide
Drug: doxorubicin hydrochloride
Drug: thalidomide
Procedure: adjuvant therapy
Procedure: conventional surgery
Procedure: neoadjuvant therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as cisplatin and doxorubicin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells. Thalidomide may stop the growth of liver cancer by blocking blood flow to the tumor. Chemoembolization kills tumor cells by blocking the blood flow to the tumor and keeping chemotherapy drugs near the tumor. Giving combination chemotherapy, thalidomide, and chemoembolization before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed. Giving thalidomide together with chemotherapy after surgery may kill any remaining tumor cells and prevent the tumor from coming back.

PURPOSE: This phase II trial is studying how well giving combination chemotherapy and thalidomide together with chemoembolization works in treating younger patients undergoing surgery for newly diagnosed liver cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the event-free and overall survival of younger patients undergoing surgery for newly diagnosed, noncirrhotic hepatocellular carcinoma (HCC) treated with neoadjuvant cisplatin, doxorubicin hydrochloride, and thalidomide (PLADOTH) followed by transarterial hepatic arterial chemoembolization comprising cisplatin and doxorubicin hydrochloride and adjuvant cyclophosphamide and thalidomide.
* Determine the efficacy and tolerability of PLADOTH in patients with initially unresectable noncirrhotic HCC treated with this regimen.
* Determine the rate of complete surgical resection by encouragement of liver transplantation in the treatment strategy as a valid option for tumor removal when partial liver resection or other surgical options remain unfeasible for patients treated with this regimen.
* Determine the long-term remission and decreased relapse rates of patients treated with this regimen based on the postoperative regimen.

Secondary

* Determine the response rate of patients treated with this regimen after treatment with PLADOTH.
* Determine the short-term toxicity and feasibility of PLADOTH in patients treated with this regimen.
* Determine the efficacy and toxicity of the postoperative regimen in terms of maintenance and duration of complete remission (no more evidence of disease and normal alpha-fetoprotein, if initially elevated) in patients treated with this regimen.
* Determine whether response to PLADOTH by the RECIST criteria can be used for better monitoring of response of patients treated with this regimen.
* Determine whether the rate of fall of serum VEGF and bFGF levels during PLADOTH can be used as prognostic factors for short-term and long-term outcome in patients treated with this regimen.
* Determine the feasibility of chemoembolization in patients treated with this regimen who do not respond to PLADOTH.
* Determine which subset of tumors may benefit from an angiostatic treatment approach based on radiological, surgical, and pathological data collected from patients treated with this regimen.
* Identify possible novel factors that might influence treatment choice and disease outcome based on radiological, surgical, and pathological data collected from patients treated with this regimen.
* Determine guidelines for diagnostic, therapeutic, and follow-up management that would improve clinical care for patients treated with this regimen.

OUTLINE: This is a multicenter, nonrandomized, open-label study.

All patients undergo either tumor biopsy or resection. Patients with localized resectable tumors undergo resection. They then proceed directly to the postoperative treatment. Patients with initially unresectable tumors undergo biopsy then proceed to the pre-operative regimen.

* Pre-operative chemotherapy and thalidomide (PLADOTH): Patients receive PLADOTH comprising cisplatin IV continuously over 24 hours on day 1, doxorubicin hydrochloride IV over 1 hour on days 1 and 2 (or IV continuously over 24 hours on days 1 and 3), and oral thalidomide daily on days 1-21. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity. Patients whose tumors are deemed resectable proceed to surgery. Patients with responding disease but whose tumors remain unresectable proceed to chemoembolization or receive 2 additional courses of PLADOTH.
* Transarterial hepatic artery chemoembolization (TACE): Patients undergo TACE comprising cisplatin and doxorubicin hydrochloride administered through a catheter placed near the tumor. TACE may be repeated every 3-4 weeks for as long as disease continues to respond or until the tumor becomes resectable. Patients also receive oral thalidomide once daily during TACE. Once the tumor is deemed resectable, patients proceed to surgery.
* Surgery: Patients undergo surgical resection of the tumor. Patients undergo either partial or total hepatectomy followed by a liver transplant and lung surgery, if necessary. Patients then proceed to the postoperative treatment.
* Postoperative treatment: Beginning within 6 weeks after surgery, patients receive oral cyclophosphamide once every other day and oral thalidomide once daily for up to 1 year in the absence of disease progression or unacceptable toxicity.

Patients with metastatic disease who show disease progression at any time during treatment go off study and receive individual advice regarding further treatment based on the decision of the principal investigator.

After completion of study treatment, patients are followed periodically for 5 years.

PROJECTED ACCRUAL: A total of 47 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed hepatocellular carcinoma (HCC) family of tumors by percutaneous needle biopsy (unless primary tumor resection is attempted)

  * Newly diagnosed disease
  * No recurrent disease
  * Fibrolamellar and transitional variants
  * Noncirrhotic disease

    * If suspicious of liver cirrhosis (e.g., abnormal liver function tests and/or positive viral serology and/or radiological evidence) at diagnosis, patient must undergo biopsy of normal liver to exclude liver cirrhosis

PATIENT CHARACTERISTICS:

* Able to follow the protocol
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Life expectancy at least 3 months
* Glomerular filtration rate ≥ 75-50% of the lower limit of normal for age (≥ 60 mL/min for patients ≥ 2 years old)
* Cardiac ejection fraction ≥ 29% at baseline ECHO

PRIOR CONCURRENT THERAPY:

* No prior treatment for HCC

Max Age: 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 47 (Estimated)
Dates: Start 2005-06; Primary Completion 2009-04 (Estimated)

PRIMARY OUTCOMES:
Event-free and overall survival following tumor resection

SECONDARY OUTCOMES:
Efficacy and tolerability following course 2 and 4 of pre-operative chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Morland, MD, Study Chair — Birmingham Children's Hospital
Locations (21):
- Our Lady's Hospital for Sick Children Crumlin, Dublin, Ireland
- United Kingdom (20):
  - Birmingham Children's Hospital, Birmingham, England
  - Institute of Child Health at University of Bristol, Bristol, England
  - Addenbrooke's Hospital, Cambridge, England
  - Leeds Cancer Centre at St. James's University Hospital, Leeds, England
  - Leicester Royal Infirmary, Leicester, England
  - Royal Liverpool Children's Hospital, Alder Hey, Liverpool, England
  - Royal London Hospital, London, England
  - Great Ormond Street Hospital for Children, London, England
  - Royal Manchester Children's Hospital, Manchester, England
  - Sir James Spence Institute of Child Health at Royal Victoria Infirmary, Newcastle upon Tyne, England
  - Queen's Medical Centre, Nottingham, England
  - Oxford Radcliffe Hospital, Oxford, England
  - Children's Hospital - Sheffield, Sheffield, England
  - Southampton General Hospital, Southampton, England
  - Royal Marsden - Surrey, Sutton, England
  - Royal Belfast Hospital for Sick Children, Belfast, Northern Ireland
  - Royal Aberdeen Children's Hospital, Aberdeen, Scotland
  - Royal Hospital for Sick Children, Edinburgh, Scotland
  - Royal Hospital for Sick Children, Glasgow, Scotland
  - Childrens Hospital for Wales, Cardiff, Wales